CLINICAL TRIAL: NCT05405491
Title: Impact of a Strategy Based on the PCR Testing System on Appropriate and Targeted Antimicrobial Treatment in Immunocompromised Patients With Suspected Ventilator-associated Pneumonia or Hospital-acquired Pneumonia Requiring Mechanical Ventilation : a Randomized Controlled Unblinded Trial
Brief Title: Impact of a Strategy Based on Bacterial DNA Detection to Optimize Antibiotics in Immunocompromised Patients With Hospital-acquired Pneumonia Requiring Mechanical Ventilation
Acronym: RESPIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021_0344; 2021-A02900-41 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia, Ventilator-Associated; Pneumonia, Hospital-Acquired; Immunodeficiency
Keywords: Ventilator-associated pneumonia; Hospital-acquired pneumonia; Immunodeficiency; Antimicrobial therapy; Polymerase chain reaction (PCR)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia; Immunologic Deficiency Syndromes | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCR group (Experimental)
  Interventions: Other: PCR based strategy
- Control group (Sham Comparator)
  Interventions: Other: Standard care

INTERVENTIONS:
Other: PCR based strategy — Early adjustment of antimicrobial therapy according to the results of a multiplex PCR-based testing, used in addition to standard microbiological culture of the tracheal aspirate, in immunocompromised patients with suspected VAP or HAP requiring MV
  Arms: PCR group
Other: Standard care — Broad-spectrum antimicrobial therapy adjustment after results of standard microbiological culture of the tracheal aspirate in immunocompromised patients with suspected VAP or HAP requiring MV
  Arms: Control group

SUMMARY:
RESPIRE is a randomized, unblinded, controlled study to measure the impact of a strategy based on a PCR test on the adjustment of antimicrobial therapy in immunocompromised patients suspected with ventilator-associated or hospital-acquired pneumonia (VAP/HAP) requiring mechanical ventilation (MV) in Intensive Care Unit (ICU). The gold-standard microbiological diagnostic method for pneumonia in the ICU is based on culture identification and antimicrobial susceptibility testing. Results are obtained in several days after the initiation of empiric antimicrobial therapy, exposing patients to a potential inappropriate broad-spectrum antimicrobial treatment. We aim to measure the impact of a PCR-based strategy to improve the percentage of patients with VAP or HAP receiving targeted antimicrobial therapy 24 hours after diagnosis compared to standard care

ELIGIBILITY:
Inclusion Criteria:

* Adult immunocompromised patients hospitalized in ICU with suspected VAP or HAP requiring MV

Exclusion Criteria:

* No immunodeficiency Moribund patients (SAPS II > 90) Pregnant women Refuse to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Increase in percentage of patients with targeted antibiotics | 24 hours after the initiation of empiric antimicrobial therapy
  To determine the impact of a PCR-based strategy on the increase in percentage of patients with targeted antibiotics regimen 24 hours after starting empiric antimicrobial therapy in the experimental group compared to standard care

SECONDARY OUTCOMES:
Percentage of patients receiving appropriate anticrobial treatment | 24 hours after the initiation of empiric antimicrobial therapy
  To determine the impact of a PCR-based strategy on the percentage of patients receiving approriate antimicrobial treatment 24 hours after starting empiric antimicrobial therapy in the experimental group compared to standard care
Mechanical ventilation free days | 28 days after the initiation of empiric antimicrobial therapy
  To determine the impact of a PCR-based strategy on the amount of days alive and free from mechanical ventilation at day 28 after the initiation of empiric antimicrobial therapy in the experimental group compared to standard care
ICU Length of stay | Until 28 days after the initiation of empiric antimicrobial therapy
  To determine the impact of a PCR-based strategy on the length of stay in the Intensive Care Unit in the experimental group compared to standard care
28 days mortality | 28 days after the initiation of empiric antimicrobial therapy
  To determine the impact of a PCR-based strategy on the mortality at Day 28 after the initiation of empiric antimicrobial therapy in the experimental group compared to standard care
Incidence of ICU-acquired infections and colonization involving multidrug resistant bacteria | 28 days after the initiation of empiric antimicrobial therapy
  To determine the impact of a PCR-based strategy on the incidence of ICU-acquired infections and ICU-acquired colonization involving multidrug resistant bacteria at Day 28 after the initiation of empiric antimicrobial therapy in the experimental group compared to standard care

CONTACTS AND LOCATIONS:
Overall Officials: Marion HOUARD, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Houard, Lille, France